CLINICAL TRIAL: NCT03253107
Title: Postgenome-based Systemic Discovery of Strong Biomarkers Predict Gastric Cancer Chemotherapy Response
Brief Title: Predicting Biomarker of Gastric Cancer Chemotherapy Response
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Su Youn Nam, Professor, Kyungpook National University Chilgok Hospital
Other Study IDs: KNUMC 2015-10-002-004
Record Dates: First submitted 2017-08-15; First posted 2017-08-17 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Gastric Cancer; Chemotherapy Effect; Predictive Cancer Model
Keywords: gastric cancer; RNA sequencing; chemotherapy response; miRNA sequencing
MeSH Terms: conditions — Stomach Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — RNA from gastric tissue and blood
  DNA from blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- responder in palliative chemotherapy: After initial chemotherapy, responder (complete remission, partial remission)
  Interventions: Drug: Chemotherapy
- non-responder in palliative chemotherapy: After initial chemotherapy, disease progression
  Interventions: Drug: Chemotherapy
- responder in adjuvant chemotherapy: complete cure and no recurrence at least 1 year after treatment
  Interventions: Drug: Chemotherapy
- non-responder in adjuvant chemotherapy: non-complete cure or recurrence within 1 year after treatment
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Institutinal standard chemotherapy as first line
  : XP (xeloda + cisplantin) or Xelox (xeloda+oxaliplitan) +/- Herceptin
  Other Names: XP or Xelox +/- Herceptin

SUMMARY:
* discovery and validation of biomarker predicting gastric cancer chemotherapy response

  * Analysis for expression level of mRNA using Next generation sequencing in gastric cancer tissue by chemotherapy response
  * Analysis for expression level of miRNA using Next generation sequencing in gastric cancer tissue and blood by chemotherapy response
  * Validation of mRNA and miRNA using qRT-PCR in multiple independent cohort
* Biological biomarkers-clinical factor combined prediction model of gastric cancer chemotherapy response

DETAILED DESCRIPTION:
* discovery and validation of biomarker predicting gastric cancer chemotherapy response

  * Analysis for expression level of mRNA in fresh frozen gastric cancer tissue by chemotherapy response (A) method of mRNA expression measurement: RNA sequencing (B) study group Palliative chemotherapy (inoperable patients)

    * institutional primary Chemotherapy regimen (XP or Xelox)

      1. response group
      2. progression group

         Post-OP adjuvant chemotherapy
    * institutional primary Chemotherapy regimen

      1. complete response group
      2. non-responder group

      <!-- -->

      1. and 2) groups: age, sex, regimen matched
  * Analysis for expression level of miRNA using Next generation sequencing in gastric cancer tissue and blood by chemotherapy response (A) method of mRNA expression measurement: RNA sequencing (B) study group

    * the same patients in mRNA sequencing
  * Validation of mRNA and miRNA in multiple independent cohort method of measurement of RNA expression: qRT-PCR
* Biological biomarkers-clinical factor combined prediction model of gastric cancer chemotherapy response combination of biologic biomarker and clinical factors to predict the chemotherapy response in gastric cancer

ELIGIBILITY:
Inclusion Criteria:

* new gastric cancer patients who has scheduled to start 1st cycle of chemotherapy
* patients who agreed this study and voluntarily assigned the informed consents.

Exclusion Criteria:

* patients who refused the study.
* patients who have other cancers
* heavy alcoholics

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: <Next generation sequencing analysis> (A) palliative chemotherapy
  1. responder (n=15)
  2. progression (n=15)
  (B) adjuvant chemotherpay
  1. complete response (n=15)
  2. non-responder (n=15)
  <qRT-PCR analysis> (Experimental set) (A) palliative chemotherapy
  1. responder (n=60)
  2. progression (n=60)
  (B) adjuvant chemotherpay
  1. complete responder (n=60)
  2. non-responder (n=60)
  (Validation set) (A) palliative chemotherapy
  1. responder (n=40)
  2. progression (n=40)
  (B) adjuvant chemotherpay
  1. complete responder (n=40)
  2. non-responder (n=40)
  1. and 2) groups: age, sex, regimen matched. Therefore this study will be nested case-control study. We will enroll 800 patients and then we will matched age, sex, and regimen in each group.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2015-11-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Discovery of predicting bio-markers for gastric cancer chemotherapy response | up to 36 months
  Discovery of predicting bio-markers for gastric cancer chemotherapy response using next generation sequencing and qRT-PCR

SECONDARY OUTCOMES:
Combination prediction model for adjuvant chemotherapy response in gastric cancer | up to 5 years
  Combination prediction model of biologic biomarkers and clinical factors for the response of adjuvant chemotherapy in gastric cancer
Combination prediction model for palliative chemotherapy response in gastric cancer | up to 3 years
  Combination prediction model of biologic biomarkers and clinical factors for the response of palliative chemotherapy in gastric cancer

CONTACTS AND LOCATIONS:
Overall Officials: Su Youn Nam, MD, PhD, Principal Investigator — Kyungpook National University Medical Center
Locations (1):
- Kyungpook National University Medical Canter, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided